CLINICAL TRIAL: NCT04518332
Title: Association of Intraoperative Cerebral and Renal Tissue Oxygen Saturation With Developmental and Socioemotional Delay and Postoperative Complications After Living Donor Liver Transplantation for Children: an Observational Study.
Brief Title: Intraoperative Cerebral and Renal Tissue Oxygen Saturation and Pediatric Living Donor Liver Transplantation Prognosis.
Acronym: rSO2-LDLT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 20200808
Record Dates: First submitted 2020-08-16; First posted 2020-08-19 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Pediatric Liver Transplantation; Developmental Delay; Postoperative Complications; Socioemotional Delay
MeSH Terms: conditions — Learning Disabilities; Postoperative Complications

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This rSO2 study is a prospective clinical study. The purpose of the rSO2 study is to investigate whether there is a correlation between the intraoperative cerebral and renal tissue oxygen saturation and the incidence of developmental and socioemotional delay after living donor liver transplantation for children. This study will also investigate whether intraoperative cerebral and renal tissue oxygen saturation are related to postoperative complications.

DETAILED DESCRIPTION:
There is high incidence of developmental and socioemotional delay and postoperative complications in pediatric living donor liver transplantation patients. In this prospective observational clinical study, the investigators aim to investigate the correlation between the intraoperative cerebral and renal tissue oxygen saturation and the incidence of developmental and socioemotional delay and postoperative complications. This study will enroll patients aged from 6 to 36 months old who are scheduled for elective standard living-donor liver transplantation and have signed informed consent before the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients (6 months< the Moon's age <36 months) who will receive standard living-donor liver transplantation (LDLT) in Renji Hospital.

Exclusion Criteria:

* Forehead skin infection, A history of liver transplantation, Multivisceral transplantation, Refused to participate the study

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This study will enroll patients aged from 6 to 36 months old who are scheduled for elective standard living-donor liver transplantation and have signed informed consent before the surgery.
Sampling Method: Non-Probability Sample
Enrollment: 123 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Developmental delay | 10days
  Developmental delay will be measured using Age and Stage Questionnaire(ASQ) after surgery.
Developmental delay | 1 month
  Developmental delay will be measured using Age and Stage Questionnaire(ASQ) after surgery.
Developmental delay | 3 months
  Developmental delay will be measured using Age and Stage Questionnaire(ASQ) after surgery.
Developmental delay | 6 months
  Developmental delay will be measured using Age and Stage Questionnaire(ASQ) after surgery.
Developmental delay | 1 year
  Developmental delay will be measured using Age and Stage Questionnaire(ASQ) after surgery.
Developmental delay | 2 years
  Developmental delay will be measured using Age and Stage Questionnaire(ASQ) after surgery.
Developmental delay | 3 years
  Developmental delay will be measured using Age and Stage Questionnaire(ASQ) after surgery.
Socioemotional Delay | 10days
  Socioemotional Delay will be measured using Age and Stage Questionnaire: Social Emotional(ASQ-SE) after surgery.
Socioemotional Delay | 1 month
  Socioemotional Delay will be measured using Age and Stage Questionnaire: Social Emotional(ASQ-SE) after surgery.
Socioemotional Delay | 3 months
  Socioemotional Delay will be measured using Age and Stage Questionnaire: Social Emotional(ASQ-SE) after surgery.
Socioemotional Delay | 6 months
  Socioemotional Delay will be measured using Age and Stage Questionnaire: Social Emotional(ASQ-SE) after surgery.
Socioemotional Delay | 1 year
  Socioemotional Delay will be measured using Age and Stage Questionnaire: Social Emotional(ASQ-SE) after surgery.
Socioemotional Delay | 2 years
  Socioemotional Delay will be measured using Age and Stage Questionnaire: Social Emotional(ASQ-SE) after surgery.
Socioemotional Delay | 3 years
  Socioemotional Delay will be measured using Age and Stage Questionnaire: Social Emotional(ASQ-SE) after surgery.

SECONDARY OUTCOMES:
Postoperative complications | 30 days
  Postoperative complications including Cardiovascular system, respiratory system, digestive system, urinary system, blood system will be screened.

CONTACTS AND LOCATIONS:
Overall Officials: Weifen Yu, MD,PhD, Study Director — Renji Hospital, School of Medicine, Shanghai Jiaotong University, China
Locations (1):
- Renji Hospital, Pudong, Shanghai Municipality, China